CLINICAL TRIAL: NCT05975918
Title: The Effect of Motivational Interview Intervention for Caregivers of Individuals With Severe Mental Disorders on Psychological Distress and Coping Attitudes
Brief Title: The Effect of Motivational Interview Intervention for Caregivers of Individuals With Severe Mental Disorders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Mehtap Akkoç, Lecturer, Kocaeli University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 123456
Record Dates: First submitted 2023-06-21; First posted 2023-08-04 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-07

CONDITIONS: Caregiver; Motivational Interview; Mental Disorder
Keywords: motivational interview; coping attitudes; caregiver; Psychological Distress; severe mental disorder
MeSH Terms: conditions — Mental Disorders | interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motivational İnterview (Experimental): The participants in the experimental group will be informed about the study through pre-interviews and data (Caregiver Identifying Characteristics Form, Patient Identifying Characteristics Form, Depression, Anxiety and Stress Scale (DASS-21), Coping Attitudes Assessment Scale) will be collected through pre-tests. A motivational interview intervention consisting of a total of 6 interviews will be conducted.Then, data will be collected with posttest (Caregiver Descriptive Characteristics Form, Patient Descriptive Characteristics Form, Depression Anxiety and Stress Scale (DASS-21), Coping Attitudes Assessment Scale).
  Interventions: Behavioral: Motivational İnterview
- Control (Other): Participants in the control group will be informed about the study through pre-interviews and data (Caregiver Identifying Characteristics Form, Patient Identifying Characteristics Form, Depression, Anxiety and Stress Scale (DASS-21), Coping Attitudes Assessment Scale) will be collected through pre-tests. 2 hours of training on coping with stress and problem solving skills will be provided. Then, data will be collected with posttest (Caregiver Descriptive Characteristics Form, Patient Descriptive Characteristics Form, Depression Anxiety and Stress Scale (DASS-21), Coping Attitudes Assessment Scale).
  Interventions: Other: Psychoeducation

INTERVENTIONS:
Behavioral: Motivational İnterview — Participants in the experimental group will be informed about the study through pre-interviews and data (Caregiver Descriptive Characteristics Form, Patient Descriptive Characteristics Form, Depression Anxiety and Stress Scale (DASS-21), Coping Attitudes Assessment Scale) will be collected through pre-tests. A motivational interview intervention consisting of a total of 6 interviews will be conducted.
  Other Names: Psychoeducation
  Arms: Motivational İnterview
Other: Psychoeducation — 2 hours of training on coping with stress and problem solving skills will be provided.
  Arms: Control

SUMMARY:
Serious mental illnesses are all chronic illnesses such as schizophrenia, schizoaffective disorder, and other psychotic disorders, major depression, and bipolar disorder, which cause impaired functioning in areas such as activities of daily living, self-care, social relationships, professional and academic life, quality time, etc. These chronic illnesses are a significant source of stress for the patient and family members. With the transition to community-based practices in the care of chronic mental illnesses, t he duties of families have increased and as a result, have had significant negative effects on caregiver and family functioning.

Caregivers face many challenges and these challenges cause caregivers to experience feelings such as anxiety, stress, fear, guilt, helplessness, hopelessness, powerlessness, loss, and anger. It is understood that families are in significant need of psychosocial support interventions that will enable them to develop effective coping methods and reduce stress and anxiety.

Themotivationall Interviewing Technique is one of the methods that can be applied to the caregivers of individuals diagnosed with chronic mental illness to adapt to the situation and cope with the difficulties they experience. Motivational Interviewing does not deal with issues such as teaching new information or ensuring acceptance of the past. It focuses on the individual's current stress, anxiety and dilemmas, goals, and plans. Studies show that any intervention that will contribute to the caregiver's coping attitude and psychological distress level will also support the empowerment of the sick individual. For this purpose, the study was planned to determine the effect of motivational interviewing intervention for caregivers of individuals with serious mental disorders on psychological distress and coping attitudes.

DETAILED DESCRIPTION:
Before starting the study, approval was obtained from the Kocaeli Health and Technology University Non-Interventional Research Ethics Committee dated 2023-38 and numbered 2023-38, and institutional permission was obtained from the community mental health center where the study would be conducted.

In the calculation of the sample of the study, the power analysis based on the statistics obtained from the study titled "Psychological distress, perceived stigma, and coping among caregivers of patients with schizophrenia" was taken as "α=0.05, 1-β (Power)= 0.95 and effect size=0.77" and accordingly, it was determined that a total of 36 people should be taken, 18 people in each group. In order to meet the sampling, possible losses and parametric test assumptions, it was decided to include a total of 60 people, 30 people each in the experimental and control groups.

The randomization method (a stratified sample list (including gender, age and number of rows) will be created by a third person who is not part of the research team, and a simple random number table will be used to assign the caregivers to the experimental and control groups) will be used.

The implementation of the research will be done in two phases. Phase 1: Piloting, identification of the intervention and control groups and pretesting

* The 6-session motivational interviewing intervention, which will be finalized according to expert opinions, will be piloted and the results will be evaluated. The intervention steps that require revision will be organized and the sample selection phase will begin.
* Caregivers who meet the research criteria and agree to participate in the study will be assigned to the experimental and control groups by randomization method.
* The experimental and control groups will be informed about the study through preliminary interviews and data (Caregiver Descriptive Characteristics Form, Patient Descriptive Characteristics Form, Depression Anxiety and Stress Scale (DASS-21), Coping Attitudes Assessment Scale) will be collected through pre-tests.

Phase 2: Intervention In the study, the intervention group will receive individual interviews based on motivational interviewing techniques, while the control group will receive a one-day group psychoeducation on coping with stress and problem solving skills.

Within the scope of this research, a total of 6 sessions of motivational interviewing interventions will be provided to the caregivers in the experimental group in 45-minute sessions. Pre-tests will be completed by adding an additional session to the first session and post-tests will be completed at the end of the last session.

Quantitative data will be analyzed with SPSS 25.0 package program using descriptive statistics (frequency distribution table) and inferential statistical tests. Significance will be evaluated at p<0.05 level.

ELIGIBILITY:
Inclusion Criteria:

* Being responsible for the care of individuals receiving services from the Community Mental Health Center
* Being the patient's primary caregiver for more than 6 months
* Over 18 years of age
* No other person to whom he/she is obliged to provide care

Exclusion Criteria:

* Being a paid caregiver
* No communication barriers

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2023-10-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
reducing psychological distress | 6 weeks
  AIl participants will be pretested and the test will be repeated after 6 weeks. Depression, Anxiety, and Stress Scale (DASS-21) will be applied as the pretest-posttest. The posttest mean scores are expected to be low after the motivational interview intervention was applied to the experimental group for 6 weeks after the pretest.
  Depression, Anxiety, and Stress Scale (DASS-21) This scale is a 4-point Likert-type scale and consists of seven questions each measuring "depression, stress, and anxiety dimensions". Getting 5 points or more from the depression sub-dimension, 4 points or more from the anxiety sub-dimension, and 8 points or more from the stress sub-dimension indicates that the individual has a related problem.

SECONDARY OUTCOMES:
increasing coping attitudes | 6 weeks
  All participants will be pretested and the test will be repeated after 6 weeks. The coping Attitudes Assessment Scale will be applied as a pretest-posttest. The posttest mean scores are expected to be low after the motivational interview intervention was applied to the experimental group for 6 weeks after the pretest.
  Coping Attitudes Assessment Scale The highest score that can be obtained from the scale is 160, and the lowest score is 40. A high score on the scale means a high level of coping attitude, and a low score means a low level of coping attitude.

CONTACTS AND LOCATIONS:
Locations (1):
- Kocaeli Health and Tecnology University, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No